CLINICAL TRIAL: NCT01327781
Title: Phase I Study of Z-Endoxifen as a Hormonal Therapy for Breast Cancer
Brief Title: Z-Endoxifen Hydrochloride in Treating Patients With Metastatic or Locally Recurrent Estrogen Receptor-Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-00847; NCI-2011-00847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000696902; MC093C; 8821 (Other: Mayo Clinic in Rochester); 8821 (Other: CTEP); P30CA015083 (NIH); P50CA116201 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-08

CONDITIONS: HER2/Neu Positive; Recurrent Breast Carcinoma; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Z-endoxifen hydrochloride) (Experimental): Patients receive Z-endoxifen hydrochloride PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Endoxifen Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Endoxifen Hydrochloride — Given PO
  Other Names: Z-Endoxifen HCl; Z-Endoxifen Hydrochloride
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and the best dose of Z-endoxifen hydrochloride in treating patients with estrogen receptor-positive (ER+) breast cancer that has spread to other places in the body (metastatic) or has come back at or near the same place as the original tumor (locally recurrent). Estrogen can cause the growth of breast cancer cells. Hormone therapy using Z-endoxifen hydrochloride may fight breast cancer by blocking the use of estrogen by tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To determine either the maximum-tolerated dose (MTD) of Z-endoxifen hydrochloride or the dose level associated with endoxifen steady state concentration (Css) of at least 2 uM in women with metastatic estrogen-receptor positive (ER+) breast cancer. (Dose Escalation Cohort) II. To describe the safety profile of Z-endoxifen (Z-endoxifen hydrochloride) at each of the doses examined. (Dose Escalation Cohort) III. To evaluate changes in vision after 2 cycles of treatment. (Dose Escalation Cohort) IV. To gather preliminary data on the clinical benefit in terms of tumor response rate and progression-free survival. (Dose Escalation Cohort) V. To evaluate the changes in the frequency and severity of hot flashes after 2 cycles of treatment. (Expansion Cohort) VI. Evaluate changes in irritability scale using a validated irritability questionnaire. (Expansion Cohort) VII. To evaluate changes in markers of bone formation and absorption after 2 cycles of treatment. (Expansion Cohort) XIII. To evaluate changes in vision after 2 cycles of treatment. (Expansion Cohort).

IX. To further characterize the safety profile of Z-endoxifen. (Expansion Cohort)

SECONDARY OBJECTIVES:

I. To characterize the plasma pharmacokinetics and urinary excretion of Z-endoxifen at each of the doses examined.

II. For patients beginning in dose level 7 as well as the expansion cohorts, we will describe any changes in tumor expression of ER (both full length and truncated forms), progesterone receptor (PR), steroid receptor co-activator (SRC)1, SRC3, as well as the insulin-like growth factor receptor (IGF)1R/phosphatidylinositol 3 kinase (PI3K)/v-akt Murine Thymoma Viral Oncogene Homolog 1 (AKT)/mammalian target of rapamycin (mTOR) pathway and proliferation-related Ki-67 antigen (Ki67) after 1 cycle of treatment (approximately 28 days).

III. To determine the frequency of estrogen receptor 1 (ESR1) mutations and the presence of antitumor activity (response rate and progression free survival [PFS]) in all patients whose tumors harbor ESR1 alterations.

IV. To determine whether the ESR1 mutations identified in pre-treatment tumor biopsies can be detected in matched plasma cell free deoxyribonucleic acid (DNA) from the same patients.

OUTLINE: This is a dose-escalation study followed by an expansion cohort study.

Patients receive Z-endoxifen hydrochloride orally (PO) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of metastatic or locally recurrent breast cancer
* ER positive defined as > 1% nuclear staining on the biopsy that was obtained at the confirmation of metastatic or locally recurrent disease
* Lesion type of either evaluable or measurable disease
* Pre- or post-menopausal female
* For the expansion cohorts: tumor that is accessible for biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Life expectancy > 16 weeks
* Capable of understanding investigational nature, potential risks and benefits of the study and able to provide written informed consent
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelet count >= 75,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (< 5 x institutional ULN if liver function test [LFT] elevations due to liver metastases)
* Creatinine =< 1.5 x institutional ULN
* Women with human epidermal growth factor (HER)-2 positive disease must have received and progressed on at least one prior anti-HER-2 directed regimen (trastuzumab, lapatinib) for their metastatic disease

  * For dose escalation cohort:

    * Any number of prior systematic therapy regimens is allowed

      * NOTE: prior systematic therapy in the adjuvant setting is not required
    * At least one prior hormone containing regimen in the metastatic setting (tamoxifen if pre-menopausal; aromatase inhibitor if post-menopausal)

      * NOTE: exception: patients that fail (defined as the development of metastatic disease while receiving an adjuvant hormone containing regimen of tamoxifen for premenopausal and aromatase inhibitor for postmenopausal) are eligible and not required to receive additional hormonal containing regimens prior to enrollment
    * At least one prior chemotherapy containing regimen in adjuvant and/or metastatic setting
  * For the expansion cohort(s):

    * At least one prior hormone containing regimen in the metastatic setting (tamoxifen if pre-menopausal; aromatase inhibitor if post-menopausal)

      * NOTE: exception: patients that fail (defined as the development of metastatic disease while receiving an adjuvant hormone containing regimen of tamoxifen for premenopausal and aromatase inhibitor for postmenopausal) are eligible and not required to receive additional hormonal containing regimens prior to enrollment
    * NOTE: a prior hormone containing regimen in the adjuvant setting is not required; a hormonal regimen containing everolimus is allowed
    * Either 1 or 2 prior chemotherapy regimens are allowed but not required such that both are in the metastatic setting or one is in the adjuvant setting and one in the metastatic setting (note, an anthracycline and taxane based regimen delivered in the adjuvant setting would be considered one regimen)
* Willingness to return to Mayo Clinic Rochester, Arizona, or Florida during treatment phase of the trial
* Dose Escalation cohort only:

  * Mandatory Translational Research Components

    * Willingness to provide biologic specimens (blood and urine)
  * Dose Escalation cohorts beginning at 160 mg/day: Mandatory Translational Research Components

    * Willingness to provide biologic specimens (tissue)
  * Dose Expansion cohort(s):

    * Mandatory Translational Research Components

      * Willingness to provide biologic specimens (blood, tissue and urine)
    * Note: The goals of this study include assessment of the biologic effects on surrogate markers of Z-endoxifen and therefore, are contingent upon availability of the biologic specimens
* Women of childbearing potential only: negative serum pregnancy test done =< 48 hours prior to registration
* Capable of swallowing 20-mg capsules

Exclusion Criteria:

* Any of the following therapies prior to registration:

  * Chemotherapy =< 3 weeks
  * Immunotherapy =< 3 weeks
  * Biologic therapy =< 3 weeks
  * Hormonal therapy =< 3 weeks
  * Monoclonal antibodies =< 3 weeks
  * Radiation therapy =< 3 weeks
  * Anti-Her-2 directed therapy =< 3 weeks
* Prior endoxifen therapy
* Prior history of:

  * Stroke =< 6 months prior to registration
  * Seizures =< 3 months prior to registration
  * Deep vein thrombosis (DVT) or pulmonary embolism (PE) =< 12 months prior to registration
  * Two or more episodes of DVT and/or PE =< 5 years prior to registration
  * Crystalline retinopathy
  * Abnormal uterine bleeding =< 1 year prior to registration
* Personal history of coagulopathy
* Active DVT and/or PE requiring anti-coagulant therapy

  * Patients who are on anti-coagulant therapy for maintenance are eligible as long as the DVT and/or PE was > 12 months prior to enrollment and there is no evidence for active thrombosis (either DVT or PE)
* Clinically symptomatic cataracts requiring imminent surgery

  * Note: patients that have cataracts that do not require surgery are eligible
* Other invasive malignancy that has been diagnosed or has recurred < 2 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Any co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment; EXCEPTION: neuropathies - if grade 2 neuropathies have been stable for at least 3 months since completion of prior treatment patient is eligible
* Tumors involving the spinal cord or heart
* Uncontrolled brain metastases

  * Note: brain metastases are not permitted on study unless the metastases have been treated by surgery or radiotherapy, and the patient has been neurologically stable and off steroids for >= 12 weeks
* Plans to begin bisphosphonates or denosumab after registration or began a bisphosphonate or denosumab regimen < 90 days before registration

  * Note: patients on a stable dose of bisphosphonates or denosumab for > 90 days prior to registration are eligible
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy or anti HER2 therapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03-25 (Actual); Primary Completion 2017-03-05 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
MTD defined as the highest dose level where at most 1 of 6 patients develops a dose limiting toxicity and 2 or more of the 3-6 patients treated at the next higher dose level develop a dose limiting toxicity | 28 days
  Assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. The maximum grade of each type of toxicity will be recorded for each patient. For each toxicity reported by dose level, the percentage of patients developing any degree of that toxicity as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.

SECONDARY OUTCOMES:
Progression-free survival | From study entry to the documentation of disease progression, assessed up to 3 months
Overall survival | From study entry to death due to any cause, assessed up to 3 months
Change in hot flash scores graded using a hot flash diary and the hot flash interference scale | Baseline to day 28
  The number and severity of hot flashes will be examined. Times series plots of hot flash scores will be constructed to visually assess changes across time within a dose level and between dose levels. In particular, for each expansion dose level, a 90% confidence interval will be constructed for the proportion of patients whose hot flash scores increase at least 2 fold from baseline after one course of treatment.

OTHER OUTCOMES:
Change in tumor expression levels of SRC3 | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of SRC1 | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of IGF1R | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of PI3K | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of AKT | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of mTOR | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of phosphorylated ribosomal protein S6 kinase kinase | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of epidermal growth factor receptor | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of HER2 | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of p42/p44 mitogen-activated protein kinase | Baseline up to day 28
  A grid (similar to a heat map) will be constructed where columns represent the proteins and the rows represent individual patients. This grid will be visual inspected for differences between expansion dose levels as well as tendencies of protein level shifts than seem to behave similarly.
Change in tumor expression levels of Ki-67 | Baseline up to day 56
  For Ki-67 by expansion dose level, a 90% binomial confidence interval for the mean change in the percentage of positive cells after 2 courses of treatment from pre-Z-endoxifen treatment levels will be determined. Also, Spearman rank correlation coefficients will be used to examine the strength of the association between the change in ER positivity, PR positivity, and Ki-67 positivity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Goetz, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota